CLINICAL TRIAL: NCT01183598
Title: Provision of Tocilizumab for Patients With Multicentric Castleman's Disease Who Have Demonstrated Benefit From Previous Tocilizumab Treatment
Brief Title: A Study to Provide RoActemra/Actemra (Tocilzumab) to Patients With Multicentric Castleman's Disease Who Demonstrated Benefit From Previous RoActemra/Actemra Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA19847
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Castleman's Disease
MeSH Terms: conditions — Castleman Disease | interventions — tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — maintenance dose

SUMMARY:
This open-label, single center study will provide RoActemra/Actemra (tocilizumab) to a maximum of 4 patients with Multicentric Castelman's Disease who have demonstrated benefit from RoActemra/Actemra in study MRA004US (Chugai Pharma USA) without major toxicities or significant adverse events. Patients will receive their most effective maintenance dose until disease progression or significant toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Evidence of improvement of one or more clinical benefit criteria with acceptable tolerability to RoActemra/Actemra in Protocol MRA001US, maintained clinical benefit in MRA004US, and completion of MRA004US
* Life expectancy > 12 weeks
* Zubrod performance status </= 3

Exclusion Criteria:

* Serious toxicity including anaphylactic reactions to tocilizumab during the MRA004US trial
* Any treatment for Multicentric Castleman's Disease except for corticosteroids within 2 weeks prior to Day 1
* Active infection requiring iv antibiotics for > 1 month and not resolving at least 1 week prior to Day 1; iv antibiotics prophylaxis for infections of implanted venous access portals is allowed
* Active viral infection within 28 days prior to Day 1
* Treatment with any investigational agent other than RoActemra/Actemra within 30 days prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Efficacy: Maintenance of hemoglobin >/=10.5 g/dL, of Zubrod Performance Status, and of improvement in fatigue and anorexia as per National Cancer Institute Common Toxicity Criteria (NCI CTC) scales | until disease progression or significant toxicity occurs
Safety: Adverse events, laboratory parameters, vital signs, electrocardiograms, chest X-rays | up to 90 days after discontinuation of treatment
Provision of tocilizumab for treatment of Multicentric Castleman's Disease to patients with evidence of clinical benefit in response to tocilizumab | until disease progression or significant toxicity occurs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Little Rock, Arkansas, United States